CLINICAL TRIAL: NCT04769960
Title: A Pilot Safety Study for Performing MRI in Patients Who Have Breast Tissue Expanders
Brief Title: Study of the Safety of MRI Scans in People Who Have Breast Tissue Expanders After Mastectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-055
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Adenocarcinoma
Keywords: breast tissue expander; breast cancer; mastectomy; 21-055; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with breast tissue expanders: Participants with breast tissue expanders that require an MRI for clinical purposes are eligible for this study.
  Interventions: Diagnostic Test: MRI Studies; Behavioral: Patient Reported Outcomes

INTERVENTIONS:
Diagnostic Test: MRI Studies — MRI scans will be performed on a 1.5T MRI scanner. Department of Radiology MRI SafetyGuidelines will be followed except regarding breast tissue expanders. Conventional MRIstudies will be performed using the standard of care clinical sequences.
Behavioral: Patient Reported Outcomes — Participants will fill out questionnaires before, immediately after, and approximately 3 months following the MRI examination +/- 1 month to evaluate for any pain or perceived changes with the breast tissue expander. The first questionnaire will obtain background participants information as well as establish a baseline pain level, the second questionnaire will evaluate any changes in pain after undergoing the MRI examination, and the last questionnaire will evaluate long term changes in pain. The patient reported outcome questionnaire will be optional at 3 months post-MRI +/-1 month.

SUMMARY:
The purpose of this study is to find out whether it is safe to perform MRI scans in people who have breast tissue expanders in place.

ELIGIBILITY:
Patients with breast tissue expanders that require an MRI for clinical purposes are eligible for this study. Patients must provide an implant card or surgical report indicated the exact make and model of their implanted tissue expander. Breast tissue expanders marked as "MRI unsafe" will be allowed with exceptions as described in the Participant exclusion criteria. While all types of MRI will be included in this study, including breast MRI, we anticipate that most of the MRI examinations ordered will evaluate the brain or spine for detecting or following metastasis.

Inclusion Criteria:

* Patient ≥ 18 years old on day of signing informed consent
* Has a breast tissue expander implanted > 28 days ago
* Patients must provide an implant card or surgical report indicated the exact make and model of their implanted tissue expander

Exclusion Criteria:

* Patients with AeroForm Tissue Expanders (manufactured by AirXpanders)
* Anyone who would normally be excluded from undergoing an MRI examination as per the Memorial Hospital for Cancer and Allied Diseases screening policy in the MRI Safety Policy (https://one.mskcc.org/sites/pub/ehs/Policies/ECSE-2009.pdf), aside from having a breast tissue expander
* Patients who are reportedly pregnant, who have a positive urine or serum pregnancy test at the time of imaging, or for which pregnancy cannot be ruled out.
* Patients who are unable to tolerate, comply or complete the MRI exam due to claustrophobia, anxiety, known psychiatric or substance abuse disorder, age, frailty, or medical instability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2026-02-19 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Safety of MRI scans for patients with breast tissue expanders | 2 years
  Our first aim is to assess the safety of imaging patients with breast tissue expanders in the MRI. Among the 50 MRI scans, if we can successfully complete at least 50, meaning that there are no issues of burning, heating, or pain in the region of the breast tissue expander that prevents the completion of the MRI, then we will declare the imaging safe and worthy of further investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Meng, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org